CLINICAL TRIAL: NCT04226209
Title: Effect of Physiotherapeutic Scoliosis Specific Exercises on Plantar Pressure Distribution and Balance in Adolescent Idiopathic Scoliosis
Brief Title: Effect of PSSE on Plantar Pressure Distribution and Balance in Scoliosis
Acronym: PSSE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Istanbul University - Cerrahpasa (Other)
Collaborators: Istanbul University (Other)
Responsible Party: Principal Investigator, Ayse Zengin Alpozgen, Asst. Prof., Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: 52010
Record Dates: First submitted 2020-01-09; First posted 2020-01-13 (Actual); Last update posted 2022-08-04 (Actual); Status verified 2022-08

CONDITIONS: Scoliosis; Adolescence; Physiotherapy; Exercise; Balance
Keywords: scoliosis; PSSE; balance; plantar pressure
MeSH Terms: conditions — Scoliosis; Motor Activity

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PSSE (Experimental): Physiotherapeutic Scoliosis-Specific Exercises PSSE group will receive corrective exercise for scoliosis
  Interventions: Other: PSSE
- Control (No Intervention): Control group will be taken to the queue list.

INTERVENTIONS:
Other: PSSE — Physiotherapeutic Scoliosis-Specific Exercises (PSSE) group will receive exercise for 30-40 mins in a day, twice in a week, totally 8 weeks and 16 hours. Control group will be taught the basic elements of corrective exercises and want them to do the practising during 8 weeks at home.
  Other Names: Control
  Arms: PSSE

SUMMARY:
The main aim of the study is to investigate the effect of Physiotherapeutic Scoliosis-Specific Exercises (PSSE) on Plantar Pressure Distribution and Balance in Adolescent Idiopathic Scoliosis (AIS). Twenty-four patients with AIS will randomly allocated to two groups. 'Schroth' exercises will apply to the PSSE group for 8 weeks (16 sessions). The control group will teach basic elements. Patients' maintenance of posture during both static and dynamic conditions (Biodex Balance System SD), distribution of foot pressure (Baropedometric Platform), foot posture (Foot Posture Index), frontal-sagittal plan posture (PostureScreen Mobile Application), body symmetry (Anterior Trunk Asymmetry Index and Posterior Trunk Asymmetry Index), deformity perception (The Walter Reed Visual Assessment Scale), quality of life (Pediatric Quality of Life Scale and SRS-22), spinal pain (Visual Analogue Scale) will assess at the first session and at the end of 8 weeks.

DETAILED DESCRIPTION:
Scoliosis is a complex 3-dimensional deformity of the spine characterized by rotation of the vertebra at least 10 degrees lateral deviation and a decrease in the normal kyphotic curvature of the spine. Although the etiology of adolescent idiopathic scoliosis (AIS) is unknown, it is the most common type of scoliosis that occurs in the period from the age of 10 until the skeletal development is completed.

It is reported in the literature that AIS is associated with balance dysfunction, vestibular system defect, proprioceptive disorder, and brain stem dysfunction. In visual, vestibular and somatosensorial systems responsible for postural control, central integration and motor response may be impaired in adolescent idiopathic scoliosis. It was also reported that the foot position and center of pressure was changed.

Postural stability can also be defined as maintaining an upright posture during standing. Different spinal deformities, such as scoliosis, can affect postural stability during upright and equilibrium activities. It has been reported that balance control problems seen in patients with AIS result from the relationship between body shape and body segments. Furthermore, lateral stability of these patients was found to be more inadequate when compared to their healthy counterparts.

Schroth method is a highly effective exercise method in adolescent idiopathic scoliosis. This method mainly focuses on the 3-dimensional scoliotic curvature formed by the combination of lateral, frontal and rotational deviation and tries to normalize the curvature of the spine by combining this curvature with stretching, strengthening and breathing exercises. It is seen that the 3D Schroth exercise method has a high effect on strength and chest expansion and also has an effect on Cobb angle, asymmetry, daily living activity, balance, vital capacity, pulmonary function and foot pressure.There are also studies showing that body weight transfer in AIS changes according to the level and shape of scoliotic curvature. However, the study investigating the effect of Schroth 3D exercises on changing body statics is quite limited and only one study found that Schroth exercises were more effective in weight distribution than Pilates exercises.

ELIGIBILITY:
Inclusion Criteria:

* To have diagnosis of Adolescence Idiopathic Scoliosis
* To be in between 10-17 years
* To be the Cobb angle which determined in Anteroposterior graphy as between 10-45 degree
* To not having any other exercise attitude about scoliosis before.

Exclusion Criteria:

* Spinal surgery or tumor history
* Accompanying mental, rheumatologic, neuromuscular, cardiovascular, pulmonary disease history
* Vision and / or hearing loss
* Disease history related to balance and vestibular system
* Injury or involvement of the lower extremities that may affect balance

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
Biodex Balance System SD | 8 week
  It is a multi-axial device used to measure an individual's maintenance of posture during both static and dynamic conditions. a)Test for static conditions: the participant were instructed to shift their weight to move a cursor toward each red, blinking target as displayed on the screen as quickly and with as much accuracy as possible. If a participant were to score a 100%, this would suggest that the individual moved in a precise and straight line to each target; higher percentage thus reflected better performance. b)Test for dynamic conditions: (1) Eyes Open, Firm Surface, (2) Eyes Closed, Firm Surface, (3) Eyes Open, Foam Surface, and (4) Eyes Closed, Foam Surface. For each of the four conditions, each participant was instructed to stand as still as they possibly could for the entire 30 seconds.The Overall Sway Index was recorded. Higher scores on the stability indices demonstrate a greater amount of postural sway or variability during that particular condition.
Baropedometric Platform | 8 week
  It allows for the analysis of the distribution of foot pressure on the ground. The platform consists of three elements and it is connected to a computer, where the transmitted data is saved and analyzed. During the test procedure, the following results could obtain: (a) average maximum loads [gr/cm2], (b) average loads [gr/cm2], (c) average foot area [cm2] and (d) right and left foot load distribution [%].
Foot Posture Index (FPI-6) | 8 week
  Foot Posture Index was used to assess the foot posture during full weight bearing. Six sub-measurements were performed, rated from +2 (highly pronated) to -2 (highly supinated) and summed up to an overall score. The sub-measurements consisted of the talar head palpation, supra and infra lateral malleolar curvature, calcaneal frontal plane position, prominence of the region of the talonavicular joint, congruence of the medial longitudinal arch and abduction/adduction of the forefoot on the rear foot. If the overall score was positive it indicated a pronated foot posture compared to a negative score, indicating a supinated foot.
Adams forward bending test | 8 week
  The subjects were in the standing position and both feet were given equal weight; cases are asked to lean forward. The measurement can be combined with a scoliometer. The scoliometer is placed parallel to the ground and measured between T1 and L5. During the measurement, care is taken that the body is parallel to the ground and the arms are loose. Baseline Scoliometer will be used for evaluations. Decreased degree is considered to be improvement.

SECONDARY OUTCOMES:
Frontal-sagittal plan posture evaluation | 8 week
  "PostureScreen Mobile" Application: Frontal and sagittal plan posture evaluation will be calculated by marking the reference points on the anterior, posterior and lateral photographs of the patient in "PostureScreen Mobile" application. The total displacement values in the anterior, posterior and lateral directions for postural impairment will be noted in "cm". Decreasing the total displacement values is considered as an improvement in postural parameters.
Body Symmetry | 8 week
  Anterior Trunk Asymmetry Index (ATSI):
  It is defined as the sum of the six indices determined on the patient's anterior photo: three frontal plane asymmetry indices (stern notch, axilla folds and waist lines) and three frontal plane plane height difference indices (acromions, axilla folds and waist lines). The Anterior Trunk Asymmetry Index score is calculated by placing the indices in the formula. The Anterior Trunk Asymmetry Index score, which represents full symmetry, is '0' and the increase in score indicates increased trunk asymmetry.
Body Symmetry | 8 week
  Posterior Trunk Asymmetry Index (POTSI):
  The Posterior Trunk Asymmetry Index parameter is defined as the sum of the six indices: the three frontal plane asymmetry index (C7, axilla folds and waist lines) and the three frontal plane height difference index (acromions, axilla folds and waist lines). The Posterior Trunk Asymmetry Index score is calculated by placing the indices on the posterior photo of the patient. The Posterior Trunk Asymmetry Index score, which represents full symmetry, is '0' and the increase in score indicates increased trunk asymmetry.
Deformity perception assessment | 8 week
  The Walter Reed Visual Assessment Scale (WRVAS):
  It is designed to understand the visual change caused by scoliosis and evaluates deformity under 7 headings. There are 5 different pictures that show different degrees of deformity. Each deformity is scored from 1 to 5; "1" is the best, "5" is the worst. The total score is obtained by summing the scores from all titles and dividing them by 7. The score ranges from 1 to 5, and a higher total score means that the perceived deformity is worse.
Health-related quality of life assessment | 8 week
  Pediatric Quality of Life Inventory:
  This inventory consists of two forms: child and family. Both forms included physical functions (8 items), emotional functions (5 items), social functions (5 items) and school functions (5 items). Scoring is done between 0-5 for each question. The total score of the inventory ranges between 0-100 points. The higher the score represents better the health-related quality of life.
Quality of life assessment for scoliosis: | 8 week
  Scoliosis Research Society-22 Questionnaire (SRS-22)
  Scoliosis Research Society-22 Questionnaire (SRS-22):
  The questionnaire assesses five domains: function, pain, personal image, mental health (five questions each) and treatment satisfaction (two questions). Each question is scored between 1 (worst) and 5 (best). In the interrogation whose total score ranged from 22 to 111, the high score indicates that the quality of life for scoliosis is better.
Spinal pain assessment | 8 week
  Visual Analogue Scale (VAS):
  It is used to quantify the pain intensity of patients. The condition that there is no pain is expressed as 0, and the condition that there is too much pain to be tolerated is expressed as 10.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University Cerrahpasa, Faculty of Health Science, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided